CLINICAL TRIAL: NCT06869356
Title: Expanded Indications of Endoscopic Submucosal Dissection for Early Gastric Cancer in China: a Multicenter, Ambispective, Observational, Open-cohort Study
Brief Title: Expanded Indications of Endoscopic Submucosal Dissection for Early Gastric Cancer in China
Status: Completed | Type: Observational
Sponsor: Beijing Friendship Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: ChiCTR1800016084
Record Dates: First submitted 2025-01-21; First posted 2025-03-11 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2018-05

CONDITIONS: Gastric Cancer Stage
Keywords: Expanded indications for ESD; Lymph node metastasis; Staging diagnosis scheme; Chinese population
MeSH Terms: conditions — Lymphatic Metastasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- D2 gastrectomy: Under the requirement of the guideline for laparoscopic gastrectomy for gastric cancer (2016 edition), laparoscopic radical gastrectomy is performed in patients.
  Interventions: Procedure: D2 gastrectomy

INTERVENTIONS:
Procedure: D2 gastrectomy — Under the requirement of the guideline for laparoscopic gastrectomy for gastric cancer (2016 edition), laparoscopic radical gastrectomy is performed in patients.

SUMMARY:
Background: The main treatment methods for early gastric cancer (EGC) include endoscopic submucosal dissection (ESD) and radical gastrectomy. However, appropriate treatment for patients who exceed the absolute indications for ESD remains unestablished. In China, evidence-based medicine for the expanding indications of ESD and accurate diagnostic staging for EGC patients are lacking. Thus, clinical studies involving Chinese patients with EGC are necessary to select appropriate treatment options and promote China's expanded indications for ESD and diagnostic staging scheme.

Methods: This is a multicenter, ambispective, observational, open-cohort study that is expected to enroll 554 patients with EGC. The study was launched in May 2018 and is scheduled to end in March 2022. All enrolled patients should meet the inclusion criteria. Case report forms and electronic data capture systems are used to obtain clinical data, which includes demographic information, results of perioperative blood- and auxiliary examinations, surgical information, results of postoperative pathology, and the outcomes of postoperative recovery and follow-up. Patients are followed up every 6 months after surgery for a minimum of 5 years. The primary endpoint is the rate of lymph node metastasis (LNM), whereas the secondary endpoints include the following: consistency, sensitivity, and specificity of the results of preoperative examinations and postoperative pathology cut off values for LNM; logistic regression model of expanded indications for ESD; and incidence of postoperative complications within the 30-day and 5-year relapse-free survival rates.

DETAILED DESCRIPTION:
This study will explore and evaluate expanded indications for ESD that match the characteristics of the Chinese population in patients with EGC and will introduce a related staging procedure and examination scheme that is appropriate for China. Ethical approval was obtained from all participating centers. The findings are expected to be disseminated through publications or presentations and will facilitate clinical decision-making in EGC.

ELIGIBILITY:
Inclusion Criteria:

Patients aged 18-75 years (regardless of sex). Patients with tumor diameter > 30 mm, ulceration (UL)(+), and differentiated mucosal carcinoma (T1a).

Patients with tumor diameter > 30 mm and differentiated, submucosal invasion depth < 500 μm (T1b SM1).

Patients with tumor diameter ≤ 30 mm and differentiated submucosal carcinoma (T1b).

Patients with tumor diameter ≤ 20 mm, UL(-), and undifferentiated (T1a). Patients with tumor diameter > 20 mm, UL(-), and undifferentiated (T1a). Patients with tumor diameter ≤ 30 mm, UL(+), and undifferentiated (T1a). Patients with tumor diameter > 30 mm, UL(+), and undifferentiated (T1a).

Exclusion Criteria:

Patients with gastric stump cancer. Patients with recurrent gastric cancer. Patients with multiple primary malignant tumors.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study aims to explore and evaluate expanded indications for ESD that match the characteristics of the Chinese population in patients with EGC, and to introduce a staging procedure and examination scheme for EGC that is appropriate for China.
Sampling Method: Non-Probability Sample
Enrollment: 1291 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2025-01-11 (Actual)

PRIMARY OUTCOMES:
Rate of lymph node metastasis | periprocedurally

SECONDARY OUTCOMES:
Accuracy, specificity, and sensitivity of gold standards | through study completion, an average of 5 year
  Postoperative histopathology of ultrasonic gastroscopy for tumor invasion depth, abdominal and pelvic enhanced computed tomography (CT) scan for LNM, pathological biopsy for tumor differentiation, and auxiliary examination for TNM staging.
Logistic regression model | Periprocedural
  To explore the corresponding logistic regression model, postoperative histopathological examination for LNM, depth of infiltration, and degree of differentiation are evaluated in the univariate analysis. Variables with statistical significance in the univariate analysis are examined in the multivariate analysis.
Complications | Periprocedural
  Postoperative complications classified as higher than Grade II
Five-year relapse-free survival rate | through study completion, an average of 5 year
  The time interval from the date of operation to the detection of tumor recurrence within 5 years is recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Friendship hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No